CLINICAL TRIAL: NCT06564428
Title: A Cohort Study of Hereditary Ovarian Cancer Risk Prediction Models and Pathogenesis Exploration
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 000000
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-05

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample for genetic testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mutation carriers: Patients presented to our hospital with a definite pathological diagnosis of epithelial ovarian cancer, who carry suspective gene mutations or have family history of cancer.
  Interventions: Genetic: Suspective gene mutations and family history
- Control group: Patients presented to our hospital with a definite pathological diagnosis of epithelial ovarian cancer, who don't carry any suspective gene mutations and have no family history of any type of cancer.

INTERVENTIONS:
Genetic: Suspective gene mutations and family history — To observe if the patients with suspective gene mutations or family history take higher risk of suffering from ovarian cancer.
  Groups: Mutation carriers

SUMMARY:
The aim of this project is to establish a bidirectional multicenter cohort of hereditary ovarian cancer and to describe the clinicopathologic features of hereditary ovarian cancer patients in our country. The risk prediction model of ovarian cancer for Chinese was established by following-up analysis of clinical and pathological information, genetic test results and detailed family history, to predict the risk of cancer in first-degree relatives of carriers of pathogenic/suspected pathogenic mutations, and to guide the intervention management of high-risk population of cancer.

The study will identify novel tumor-causing mutations/predisposing genes by gene sequencing in a special family with hereditary tumor.

DETAILED DESCRIPTION:
About 10%-20% of ovarian cancers have familial aggregation, suggesting that it may be hereditary ovarian cancer. Exploring a genetic ovarian cancer risk prediction model suitable for Chinese people will help quantify the risk of cancer in high risk groups and guide preventive interventions. The clinicopathology, gene mutation and family history of hereditary ovarian cancer need to be deeply analyzed, and the relevant research is still in the initial stage in China. At the same time, in a small number of ovarian cancer families with obvious familial aggregation, genetic testing failed to detect known pathogenic/possible pathogenic mutations in the germ line, suggesting that there may be a new pathogenic mechanism that needs further study.

Based on the above clinical issues, this project intends to establish a prospective multicenter cohort of hereditary ovarian cancer. To describe the clinicopathological and genetic mutation characteristics of hereditary ovarian cancer patients in China, and guide the individualized diagnosis and treatment of patients. Through follow-up analysis of clinicopathological information, gene mutation characteristics, detailed family history and other factors, a suitable ovarian cancer risk prediction model was established and preliminarily verified to guide the intervention management of high-risk groups. Special genetic ovarian cancer families or early-onset ovarian cancer cases were collected, and new tumor-causing mutations/susceptibility genes were explored through gene sequencing analysis, and functional verification and preliminary mechanism studies were conducted.

Relying on the National Clinical Research Center for Obstetrics and Gynecology, the research team has been engaged in the clinical diagnosis, treatment and scientific research of gynecological malignant tumors for a long time. In China, the gynecological tumor genetic consultation clinic was established earlier, and there are mature platforms for diagnosis, treatment and genetic blocking of hereditary ovarian cancer. Our research group has initially established a genetic ovarian cancer cohort in our hospital, which has included more than 1000 cases of patients with epithelial ovarian cancer and their families who have received surgical treatment in our hospital since 2016. In September 2022, it led the establishment of a multi-center gynecological tumor genetic diagnosis and treatment platform, with 11 sub-centers across the country working together to focus on the diagnosis, treatment and research of hereditary gynecological tumors.

The development of this project will establish the ovarian cancer risk prediction model suitable for Chinese people for the first time, and guide the prevention and intervention of high-risk groups. Through special genetic ovarian cancer family mining, to explore the new pathogenic mechanism of ovarian cancer, to guide the early diagnosis of hereditary ovarian cancer; At the same time, it will promote the individualized and accurate diagnosis and treatment of hereditary ovarian cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Epithelial ovarian cancer
* ≥18 years
* The pathological diagnosis was clear
* The genetic test showed germ line pathogenic/suspected pathogenic mutations (for mutation interpretation, refer to the American ACMG Classification Standards and Guidelines for Genetic Variation)

Exclusion Criteria:

* Non-epithelial ovarian cancer was confirmed by pathology
* No genetic test has been performed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese female population of different regions and different ages.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The clinicopathological features and gene mutation characteristics of hereditary ovarian cancer | 2024-2026
  * personal history (age, BMI, oral contraceptive use, hormone replacement therapy use, tubal ligation)
    * menstrual marriage and childbearing history (whether or not menopause, menopausal age, menarche age, the number of births)
      * personal history of tumor (history of malignant tumor, tumor type, pathological type, tumor stage, age of onset) ④family history of cancer (family history of cancer or not, number/person of cancer in first/second/third degree relatives, relationship with patients, tumor type, pathological type, tumor stage, age of onset, gene detection) ⑤results of gene detection (detection items, specimen type, mutation, mutated gene, cDNA change, amino acid change, mutation type, mutation significance)

SECONDARY OUTCOMES:
Newly diagnosed ovarian cancer in a first-degree relative | 2024-2026
  The pathological diagnosis was epithelial ovarian cancer

CONTACTS AND LOCATIONS:
Overall Officials: Hongyan Guo, Doctor, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lheureux S, Gourley C, Vergote I, Oza AM. Epithelial ovarian cancer. Lancet. 2019 Mar 23;393(10177):1240-1253. doi: 10.1016/S0140-6736(18)32552-2. PMID 30910306
- [Background] Nielsen FC, van Overeem Hansen T, Sorensen CS. Hereditary breast and ovarian cancer: new genes in confined pathways. Nat Rev Cancer. 2016 Sep;16(9):599-612. doi: 10.1038/nrc.2016.72. Epub 2016 Aug 12. PMID 27515922
- [Background] Yoshida R. Hereditary breast and ovarian cancer (HBOC): review of its molecular characteristics, screening, treatment, and prognosis. Breast Cancer. 2021 Nov;28(6):1167-1180. doi: 10.1007/s12282-020-01148-2. Epub 2020 Aug 29. PMID 32862296
- [Background] Lynch HT, Snyder CL, Shaw TG, Heinen CD, Hitchins MP. Milestones of Lynch syndrome: 1895-2015. Nat Rev Cancer. 2015 Mar;15(3):181-94. doi: 10.1038/nrc3878. Epub 2015 Feb 12. PMID 25673086
- [Background] US Preventive Services Task Force; Owens DK, Davidson KW, Krist AH, Barry MJ, Cabana M, Caughey AB, Doubeni CA, Epling JW Jr, Kubik M, Landefeld CS, Mangione CM, Pbert L, Silverstein M, Simon MA, Tseng CW, Wong JB. Risk Assessment, Genetic Counseling, and Genetic Testing for BRCA-Related Cancer: US Preventive Services Task Force Recommendation Statement. JAMA. 2019 Aug 20;322(7):652-665. doi: 10.1001/jama.2019.10987. PMID 31429903
- [Background] Gilpin CA, Carson N, Hunter AG. A preliminary validation of a family history assessment form to select women at risk for breast or ovarian cancer for referral to a genetics center. Clin Genet. 2000 Oct;58(4):299-308. doi: 10.1034/j.1399-0004.2000.580408.x. PMID 11076055
- [Background] Evans DG, Eccles DM, Rahman N, Young K, Bulman M, Amir E, Shenton A, Howell A, Lalloo F. A new scoring system for the chances of identifying a BRCA1/2 mutation outperforms existing models including BRCAPRO. J Med Genet. 2004 Jun;41(6):474-80. doi: 10.1136/jmg.2003.017996. PMID 15173236
- [Background] Bellcross CA, Lemke AA, Pape LS, Tess AL, Meisner LT. Evaluation of a breast/ovarian cancer genetics referral screening tool in a mammography population. Genet Med. 2009 Nov;11(11):783-9. doi: 10.1097/GIM.0b013e3181b9b04a. PMID 19752737
- [Background] Hoskins KF, Zwaagstra A, Ranz M. Validation of a tool for identifying women at high risk for hereditary breast cancer in population-based screening. Cancer. 2006 Oct 15;107(8):1769-76. doi: 10.1002/cncr.22202. PMID 16967460
- [Background] Ashton-Prolla P, Giacomazzi J, Schmidt AV, Roth FL, Palmero EI, Kalakun L, Aguiar ES, Moreira SM, Batassini E, Belo-Reyes V, Schuler-Faccini L, Giugliani R, Caleffi M, Camey SA. Development and validation of a simple questionnaire for the identification of hereditary breast cancer in primary care. BMC Cancer. 2009 Aug 14;9:283. doi: 10.1186/1471-2407-9-283. PMID 19682358
- [Background] Berliner JL, Cummings SA, Boldt Burnett B, Ricker CN. Risk assessment and genetic counseling for hereditary breast and ovarian cancer syndromes-Practice resource of the National Society of Genetic Counselors. J Genet Couns. 2021 Apr;30(2):342-360. doi: 10.1002/jgc4.1374. Epub 2021 Jan 7. PMID 33410258
- [Background] Berry DA, Parmigiani G, Sanchez J, Schildkraut J, Winer E. Probability of carrying a mutation of breast-ovarian cancer gene BRCA1 based on family history. J Natl Cancer Inst. 1997 Feb 5;89(3):227-38. doi: 10.1093/jnci/89.3.227. PMID 9017003
- [Background] Parmigiani G, Berry D, Aguilar O. Determining carrier probabilities for breast cancer-susceptibility genes BRCA1 and BRCA2. Am J Hum Genet. 1998 Jan;62(1):145-58. doi: 10.1086/301670. PMID 9443863
- [Background] Berry DA, Iversen ES Jr, Gudbjartsson DF, Hiller EH, Garber JE, Peshkin BN, Lerman C, Watson P, Lynch HT, Hilsenbeck SG, Rubinstein WS, Hughes KS, Parmigiani G. BRCAPRO validation, sensitivity of genetic testing of BRCA1/BRCA2, and prevalence of other breast cancer susceptibility genes. J Clin Oncol. 2002 Jun 1;20(11):2701-12. doi: 10.1200/JCO.2002.05.121. PMID 12039933
- [Background] Antoniou AC, Pharoah PD, McMullan G, Day NE, Stratton MR, Peto J, Ponder BJ, Easton DF. A comprehensive model for familial breast cancer incorporating BRCA1, BRCA2 and other genes. Br J Cancer. 2002 Jan 7;86(1):76-83. doi: 10.1038/sj.bjc.6600008. PMID 11857015
- [Background] Antoniou AC, Pharoah PP, Smith P, Easton DF. The BOADICEA model of genetic susceptibility to breast and ovarian cancer. Br J Cancer. 2004 Oct 18;91(8):1580-90. doi: 10.1038/sj.bjc.6602175. PMID 15381934
- [Background] Lee A, Mavaddat N, Cunningham A, Carver T, Ficorella L, Archer S, Walter FM, Tischkowitz M, Roberts J, Usher-Smith J, Simard J, Schmidt MK, Devilee P, Zadnik V, Jurgens H, Mouret-Fourme E, De Pauw A, Rookus M, Mooij TM, Pharoah PP, Easton DF, Antoniou AC. Enhancing the BOADICEA cancer risk prediction model to incorporate new data on RAD51C, RAD51D, BARD1 updates to tumour pathology and cancer incidence. J Med Genet. 2022 Dec;59(12):1206-1218. doi: 10.1136/jmedgenet-2022-108471. Epub 2022 Sep 26. PMID 36162851
- [Background] Dareng EO, Tyrer JP, Barnes DR, Jones MR, Yang X, Aben KKH, Adank MA, Agata S, Andrulis IL, Anton-Culver H, Antonenkova NN, Aravantinos G, Arun BK, Augustinsson A, Balmana J, Bandera EV, Barkardottir RB, Barrowdale D, Beckmann MW, Beeghly-Fadiel A, Benitez J, Bermisheva M, Bernardini MQ, Bjorge L, Black A, Bogdanova NV, Bonanni B, Borg A, Brenton JD, Budzilowska A, Butzow R, Buys SS, Cai H, Caligo MA, Campbell I, Cannioto R, Cassingham H, Chang-Claude J, Chanock SJ, Chen K, Chiew YE, Chung WK, Claes KBM, Colonna S; GEMO Study Collaborators; GC-HBOC Study Collaborators; EMBRACE Collaborators; Cook LS, Couch FJ, Daly MB, Dao F, Davies E, de la Hoya M, de Putter R, Dennis J, DePersia A, Devilee P, Diez O, Ding YC, Doherty JA, Domchek SM, Dork T, du Bois A, Durst M, Eccles DM, Eliassen HA, Engel C, Evans GD, Fasching PA, Flanagan JM, Fortner RT, Machackova E, Friedman E, Ganz PA, Garber J, Gensini F, Giles GG, Glendon G, Godwin AK, Goodman MT, Greene MH, Gronwald J; OPAL Study Group; AOCS Group; Hahnen E, Haiman CA, Hakansson N, Hamann U, Hansen TVO, Harris HR, Hartman M, Heitz F, Hildebrandt MAT, Hogdall E, Hogdall CK, Hopper JL, Huang RY, Huff C, Hulick PJ, Huntsman DG, Imyanitov EN; KConFab Investigators; HEBON Investigators; Isaacs C, Jakubowska A, James PA, Janavicius R, Jensen A, Johannsson OT, John EM, Jones ME, Kang D, Karlan BY, Karnezis A, Kelemen LE, Khusnutdinova E, Kiemeney LA, Kim BG, Kjaer SK, Komenaka I, Kupryjanczyk J, Kurian AW, Kwong A, Lambrechts D, Larson MC, Lazaro C, Le ND, Leslie G, Lester J, Lesueur F, Levine DA, Li L, Li J, Loud JT, Lu KH, Lubinski J, Mai PL, Manoukian S, Marks JR, Matsuno RK, Matsuo K, May T, McGuffog L, McLaughlin JR, McNeish IA, Mebirouk N, Menon U, Miller A, Milne RL, Minlikeeva A, Modugno F, Montagna M, Moysich KB, Munro E, Nathanson KL, Neuhausen SL, Nevanlinna H, Yie JNY, Nielsen HR, Nielsen FC, Nikitina-Zake L, Odunsi K, Offit K, Olah E, Olbrecht S, Olopade OI, Olson SH, Olsson H, Osorio A, Papi L, Park SK, Parsons MT, Pathak H, Pedersen IS, Peixoto A, Pejovic T, Perez-Segura P, Permuth JB, Peshkin B, Peterlongo P, Piskorz A, Prokofyeva D, Radice P, Rantala J, Riggan MJ, Risch HA, Rodriguez-Antona C, Ross E, Rossing MA, Runnebaum I, Sandler DP, Santamarina M, Soucy P, Schmutzler RK, Setiawan VW, Shan K, Sieh W, Simard J, Singer CF, Sokolenko AP, Song H, Southey MC, Steed H, Stoppa-Lyonnet D, Sutphen R, Swerdlow AJ, Tan YY, Teixeira MR, Teo SH, Terry KL, Terry MB; OCAC Consortium; CIMBA Consortium; Thomassen M, Thompson PJ, Thomsen LCV, Thull DL, Tischkowitz M, Titus L, Toland AE, Torres D, Trabert B, Travis R, Tung N, Tworoger SS, Valen E, van Altena AM, van der Hout AH, Van Nieuwenhuysen E, van Rensburg EJ, Vega A, Edwards DV, Vierkant RA, Wang F, Wappenschmidt B, Webb PM, Weinberg CR, Weitzel JN, Wentzensen N, White E, Whittemore AS, Winham SJ, Wolk A, Woo YL, Wu AH, Yan L, Yannoukakos D, Zavaglia KM, Zheng W, Ziogas A, Zorn KK, Kleibl Z, Easton D, Lawrenson K, DeFazio A, Sellers TA, Ramus SJ, Pearce CL, Monteiro AN, Cunningham J, Goode EL, Schildkraut JM, Berchuck A, Chenevix-Trench G, Gayther SA, Antoniou AC, Pharoah PDP. Polygenic risk modeling for prediction of epithelial ovarian cancer risk. Eur J Hum Genet. 2022 Mar;30(3):349-362. doi: 10.1038/s41431-021-00987-7. Epub 2022 Jan 14. PMID 35027648
- [Background] Daly MB, Pilarski R, Yurgelun MB, Berry MP, Buys SS, Dickson P, Domchek SM, Elkhanany A, Friedman S, Garber JE, Goggins M, Hutton ML, Khan S, Klein C, Kohlmann W, Kurian AW, Laronga C, Litton JK, Mak JS, Menendez CS, Merajver SD, Norquist BS, Offit K, Pal T, Pederson HJ, Reiser G, Shannon KM, Visvanathan K, Weitzel JN, Wick MJ, Wisinski KB, Dwyer MA, Darlow SD. NCCN Guidelines Insights: Genetic/Familial High-Risk Assessment: Breast, Ovarian, and Pancreatic, Version 1.2020. J Natl Compr Canc Netw. 2020 Apr;18(4):380-391. doi: 10.6004/jnccn.2020.0017. PMID 32259785

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-05-02): https://cdn.clinicaltrials.gov/large-docs/28/NCT06564428/Prot_SAP_ICF_001.pdf